CLINICAL TRIAL: NCT00845455
Title: Personality Type as a Predictor to Develop Depression and Reduction in Quality of Life Among Stroke Survivals.
Acronym: TPQ BDI SSQOL
Status: Completed | Type: Observational
Sponsor: d_yarnitsky (Other)
Responsible Party: Sponsor-Investigator, d_yarnitsky, MD, Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Other Study IDs: TPQStroke03CTIL
Record Dates: First submitted 2009-02-15; First posted 2009-02-18 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Stroke; Depression; Quality of Life; Personality Type
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1. Harm Avoidance: Personality type
- 2. Reward Dependence: Personality type
- 3. Novelty Seeking: Personality type

SUMMARY:
Personality type as a predictor to develop depression and reduction in quality of life among stroke survivals.

ELIGIBILITY:
Inclusion Criteria:

* any stroke,
* age 40-90,
* able to sigh informed concent,
* able to fill in the questionnaires.

Exclusion Criteria:

* non stroke,
* previous depression,
* not able to give consent or answer the questions.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke ( TIA, CVA, ICH ) patients
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Depression | 1-3 month post stroke

SECONDARY OUTCOMES:
QOL post stroke | 1-3 month post stroke

CONTACTS AND LOCATIONS:
Overall Officials: David - Yarnitsky, Prof., Principal Investigator